CLINICAL TRIAL: NCT04634318
Title: Organization of Pulmonary Rehabilitation of Post-COVID-19 Patient With Sequelae. Assessment and Therapeutic Indication of Tele-rehabilitation Versus Conventional Rehabilitation
Brief Title: Organization of Pulmonary Rehabilitation of Post-COVID-19 Patient With Sequelae (REHABCOVID)
Acronym: REHABCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-CHITS-06; 2020-A02838-31 (Other: Id-RCB)
Record Dates: First submitted 2020-11-17; First posted 2020-11-18 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-10

CONDITIONS: Covid19
Keywords: COVID19; Sequelae; Dyspnea; Exercise intolerance; Respiratory rehabilitation; Telemedicine
MeSH Terms: conditions — COVID-19; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory rehabilitation program group (RR). (Active Comparator): Post-COVID-19 patients carrying out a respiratory rehabilitation program (RR).
  Interventions: Other: Respiratory rehabilitation program (RR).
- Respiratory tele-rehabilitation program group (TRR). (Experimental): Post-COVID-19 patients carrying out a respiratory tele-rehabilitation program (TRR).
  Interventions: Other: Respiratory tele-rehabilitation program (TRR).

INTERVENTIONS:
Other: Respiratory rehabilitation program (RR). — Patients in the RR group will follow the respiratory rehabilitation program during a 4-week hospitalization in the respiratory diseases department of Renée Sabran hospital (Hyères, France).
  The program includes for each week:
  One medical consultation Four 40-min sessions of aerobic exercises on an ergocycle Four 1-hour sessions of walking in Renée Sabran Hospital's park Three 1-hour sessions of muscle strengthening exercises One 1-hour session of sophrology One 1-hour session of occupational therapy One 1-hour session of psychomotricity
  Arms: Respiratory rehabilitation program group (RR).
Other: Respiratory tele-rehabilitation program (TRR). — Patients in the TRR group will realize the 4-week respiratory tele-rehabilitation program at home. The TRR program for each week includes the same sessions as RR program. But, medical consultation, sophrology, occupational therapy, psychomotricity and muscle strengthening sessions are carried out through live videoconferences. Additionally, aerobic and walking sessions are carried out outside home. The intensity of each session will be controlled by heart rate monitor.
  Arms: Respiratory tele-rehabilitation program group (TRR).

SUMMARY:
Some patients with COVID-19 have sequelae after the acute phase of infection. These sequelae can be physical (dyspnea, exercise intolerance, abnormal fatigue) but also psychic (anxiety, depression). Systemic sequelae have also been observed in pulmonary, cardiac, hepatic, renal, nervous or immune systems. Respiratory rehabilitation (RR) is indicated in these patients to help their complete recovery without sequelae. These patients' arrival and sanitary constraints imposed by COVID-19 changed the organization of Health Care Centers (HCC). Risk of contagiousness after the acute phase of infection still exists. Consequently, patients must respect a quarantine time on their arrival in HCC and then have no contact with other HCC patients to respect the barrier rules and social distancing measures. HCC accommodation capacities are reduced and this is to the detriment of patients with chronic diseases for whom RR is essential. Certain HCCs saturation can also be responsible for a non-proposal of RR in the care pathway of patients after COVID-19. To cope with the new constraints imposed by Covid-19 pandemic, telemedicine is being developed in the affected industrial countries. Some SRH physicians are starting to offer post-COVID-19 patients the possibility of carrying out a tele-rehabilitation program (TRR). Such a telemedicine program has been validated for people with respiratory failure. It allows the patient to follow his care program without leaving his home and it does not require the visit from a health professional. In addition to reducing the inflow of post COVID-19 patients in HCC, it allows fragile patients to respect social distancing. It could also contain virus spread virus on the territory by reducing patient movements. When choosing between RR and TRR, the clinician must ask himself two questions. Is TRR as efficient as RR for post-COVID-19 patients? Is there a profile of patients for whom either method gives better results? This study proposes to evaluate both methods: a 4-week TRR program vs a conventional RR program in post COVID-19 patients with sequelae. If the hypothesis that both methods have similar effects is verified, this would allow the generalization of the prescription of TRR. The benefits will be individual with greater access to respiratory rehabilitation for post COVID-19 patients. There will also be collective public health benefits by maintaining sufficient access to HCC for patients with chronic diseases.

DETAILED DESCRIPTION:
Some COVID-19 patients have sequelae after infection acute phase. These sequelae can be physical (dyspnea, exercise intolerance, abnormal fatigue) but also psychic (anxiety, depression). Systemic sequelae have also been observed in pulmonary, cardiac, hepatic, renal, nervous or immune systems. Respiratory rehabilitation (RR) is indicated in these patients to help their complete recovery. Regional Health Agencies (ARS) have listed Health Care Centers (HCCs) that can welcome these patients. Their arrival and sanitary constraints imposed by COVID-19 changed these HCC organization. Risk of contagiousness after infection acute phase still exists. Consequently, patients must first respect a quarantine time and then have no contact with other HCC patients to respect barrier rules. HCC accommodation capacities are reduced to the detriment of patients with chronic diseases for whom RR is essential. Certain SSRs saturation can also be responsible for a non-proposal of RR to COVID-19 patients. To cope with the new constraints imposed by COVID-19, telemedicine is being developed in affected industrial countries. Some SRH physicians are starting to offer post-COVID-19 patients a tele-rehabilitation program (TRR). Such a program has been validated for people with respiratory failure. It allows a patient to follow his care program without leaving home and it does not require health professional visits. In addition to reducing post COVID-19 patient inflow in HCC, it allows fragile patients to respect social distancing and could contain virus spread on the territory by reducing patient movements. When choosing between RR and TRR, a clinician must ask himself two questions. Is TRR as efficient as RR for post-COVID-19 patients? Is there a profile of patients for whom either method gives better results? This study evaluates both methods: a 4-week TRR program vs a conventional RR program. If the hypothesis that both methods have similar effects is verified, this would allow TRR prescription generalization. Benefits will be individual with greater access to respiratory rehabilitation for post COVID-19 patients. There will also be collective benefits by maintaining sufficient SSR access for patients with chronic diseases.

This study could also help clinicians to choose the best therapeutic methods to combat post COVID-19 sequelae. Indeed, effectiveness study of rehabilitation programs according to medical, physical and psychological patient profile will define what is the most suitable post COVID-19 care method (TRR or RR) for each patient. Thus, it could help to determine the characteristics of the patients for whom a tele-rehabilitation program is indicated.

Sessions carried out in RR and TRR programs are similar. Session number is the same in both programs. They have the same goal and the same intensity. In RR program, sessions are carried out at Renée Sabran Hospital, supervised by medical staff. In TRR program, sessions are carried out at patient's home, supervised by medical staff by video-conference. Additionally, aerobic and walking sessions are carried out outside home. The intensity of each session will be controlled by heart rate monitor.

The same outcome measurements are carried out before and after both respiratory rehabilitation programs. To verify that both respiratory rehabilitation programs have similar efficiency, outcome measures will be analyzed using a 2-factor analysis of variance:

* group (TRR vs RR)
* time (before vs after respiratory rehabilitation program)

Relationship between effectiveness of both respiratory rehabilitation programs and the different characteristics of patients when programs start will be analyzed using multiple linear regression.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18 years old.
* Subjects having contracted COVID-19 as evidenced by a positive RT-PCR test and / or the presence of antibodies.
* Subjects having had a medical prescription for respiratory rehabilitation.
* Subject having the hardware and network coverage necessary to achieve a videoconference.
* Subjects with at least one of the following post-COVID-19 sequelae:

  * Dyspnea at rest or during exercise objectified by the mMRC (modified Medical Research Council) scale with a score greater than or equal to 2. (Vestbo et al, 2013)
  * Dysfunction of ventilation objectified by the Nijmegen questionnaire with a score greater than or equal to 23/64 (Van Dixhoorn and Duivenvoordent, 1985)
  * Exercise intolerance objectified by the 1min-STS according to the standards by age and sex established by Strassmann et al (2013).
  * Abnormal fatigue objectified by the MFI-20 (Multidimensional Fatigue Inventory) validated in French by Gentile et al (2003) according to the age and sex standards established by Schwarz et al (2003).
  * State of anxiety or depression objectified by the HADS (Hospital Anxiety and Depression scale) validated in French by Roberge et al (2013) according to the standards by age and sex established by Bocéréan and Ducret (2014)
* Patients covered by social security or equivalent regimen

Exclusion Criteria:

* Subjects infected again by SARS-CoV-2 during the study as evidenced by a positive RT-PCR test
* Every deterioration of patient physical or psychological state (linked for example to injury or disease) requiring rehabilitation program arrest or incapacity to perform functional tests or to answer questionnaires
* Cardio-vascular contraindications to exercise
* Instability of the respiratory state
* Neuromuscular, osteoarticular or psychiatric disease making exercise impossible
* Person presenting severe depression according to DSM-5 criteria
* Person being in the exclusion period of another research protocol at the moment of inclusion
* Person not mastering enough French language reading and understanding to be able to consent in writing to participate in the study
* Every condition which, according to investigator, might increase or compromise the person security in case of study participation
* Patient with medical history which, according to investigator, might interfere with objective assessment and study results
* Pregnant or breastfeeding women
* Patient deprived of liberty by judicial or administrative decision
* Patient under legal protection measure or not able to express his consent
* Patient not able to follow study procedures and to respect the visits during all study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Distance walked in the 6-min walk test (6 MWT). | 8 weeks
  The 6-min walk test (6 MWT) measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes (the 6MWD). (ATS Statement: Guidelines for the Six-Minute Walk Test, Am J Respir Crit Care Med, 2002)

SECONDARY OUTCOMES:
Number of repetitions performed in a 1-min Sit-to-Stand (STS) test | 8 weeks
  All 1-min STS tests are performed according to a standardized protocol by trained study staff. A standard chair is used (height 46-48 cm) with a flat seat and no armrests, stabilized against a wall. Patients are asked to sit with their legs hip-width apart and flexed to 90°, with their hands stationary on the hips without using the hands or arms to assist movement. They are instructed to stand completely straight and touch the chair with their bottom when sitting, but they need not sit fully back on the chair. Patients are asked to perform as many repetitions as possible in 1 min, and after 45 s are told "you have 15 s left until the test is over". (Crook S, et al. Eur Respir J 2017)
Dyspnea evaluated by the modified Medical Research Council (mMRC) | 8 weeks
  The mMRC dyspnea scale allows to assess degree of baseline functional disability due to dyspnea. (Vestbo J, et al. Am J Respir Crit Care Med, 2013)
Fatigue evaluated by the Multidimensional Fatigue Inventory (MFI-20) | 8 weeks
  Multidimensional Fatigue Inventory (MFI-20) is a 20-item self-report instrument which covers the following dimensions: general fatigue, physical fatigue, reduced activity, reduced motivation, and mental fatigue (Schwarz, et al. Onkologie, 2003)
Anxiety and Depression evaluated by the Hospital Anxiety and Depression Scale (HADS) | 8 weeks
  The Hospital Anxiety and Depression Scale (HADS) can be useful tools for identifying potential cases of anxiety and depression (Roberge P, et al. J Affect Disord.2013)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Vallier, MD, Study Director — Toulon University
Locations (3):
- France (3):
  - Hôpital Nord (AP-HM), Marseille, Bouches Du Rhône
  - Hôpital Renée Sabran, Hyères, Var
  - HIA Sainte Anne, Toulon, Var

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Crook S, Puhan MA, Frei A; STAND-UP and RIMTCORE study groups. The validation of the sit-to-stand test for COPD patients. Eur Respir J. 2017 Sep 20;50(3):1701506. doi: 10.1183/13993003.01506-2017. Print 2017 Sep. No abstract available. PMID 28931670
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Background] Schwarz R, Krauss O, Hinz A. Fatigue in the general population. Onkologie. 2003 Apr;26(2):140-4. doi: 10.1159/000069834. PMID 12771522
- [Background] Roberge P, Dore I, Menear M, Chartrand E, Ciampi A, Duhoux A, Fournier L. A psychometric evaluation of the French Canadian version of the Hospital Anxiety and Depression Scale in a large primary care population. J Affect Disord. 2013 May;147(1-3):171-9. doi: 10.1016/j.jad.2012.10.029. Epub 2012 Dec 4. PMID 23218249
- [Result] Vallier JM, Simon C, Bronstein A, Dumont M, Jobic A, Paleiron N, Mely L. Randomized controlled trial of home-based vs. hospital-based pulmonary rehabilitation in post COVID-19 patients. Eur J Phys Rehabil Med. 2023 Feb;59(1):103-110. doi: 10.23736/S1973-9087.22.07702-4. Epub 2023 Jan 26. PMID 36700245